CLINICAL TRIAL: NCT07230925
Title: Study of the Rate of Progression of Cerebral Ischemia in Afro-Caribbeans
Acronym: VESPERALS
Status: Not yet recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire de la Guadeloupe (Other)
Responsible Party: Sponsor
Other Study IDs: PAP_RIPH2_2025/03
Record Dates: First submitted 2025-11-14; First posted 2025-11-17 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-10

CONDITIONS: Ischemic Stroke; Cerebral Ischemia; Endovascular Treatments
Keywords: Cerebrovascular accident; Cerebral Blood Flow
MeSH Terms: conditions — Ischemic Stroke; Brain Ischemia; Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients residing in Guadeloupe: Patients residing in Guadeloupe
  Interventions: Other: No Interventions
- Patients residing in Nantes: Patients residing in Nantes
  Interventions: Other: No Interventions

INTERVENTIONS:
Other: No Interventions — No interventions

SUMMARY:
To compare the progression of cerebral ischemia from HF in Afro-Caribbean patients admitted to the CHUG to that of patients from Nantes included in the national ETIS registry.

DETAILED DESCRIPTION:
mpare the progression of cerebral ischemia of IC in Afro-Caribbean patients admitted to the CHUG with that of patients from Nantes included in the national register ETIS.

Secondary outcomes: Stroke is a sudden interruption of blood flow in the brain. Among the types of stroke, cerebral infarction is the most common (80% of cases). Cerebral infarction (CI) is a sudden disruption of brain circulation due to the occlusion of an artery by a clot. Large vessel occlusions (OLV) of the brain represent 30-40% of occlusions and are frequently associated with poor prognosis. Mechanical thrombectomy (MT) involves the extraction of the intra-arterial thrombus. Often performed in conjunction with intravenous thrombolysis (TIV), it has become the preferred treatment for OLV. However, not all patients with OLV are eligible for TM. It is recognized that for the same occlusion site, the rate of progression of HF varies from individual to individual. There are two categories of patients: the "fast progressor" and the "slow progressor". Patients referred to as "fast progressor" have a higher volume CI than "slow progressors" for the same time delay between onset of symptoms and imaging. The "fast progressor" profile is usually associated with an unfavourable functional prognosis. In the study by Rocha et al (ref. n°8), assessing the prevalence and distribution of ischemic volume progression rate in patients with OLV; 58% of patients had ischemic volume 30 mL and 72% had ischemic volume 70 mL within 24 hours after the onset of stroke. These patients were characterized as "slow progressors".

In 2022, a retrospective preliminary study was carried out at the Guadeloupe University Hospital and allowed for a comparison of patients treated within the institution with those of patients from the ETIS Register recording thrombectomies performed nationally. The comparison between the two populations shows that patients who have suffered a stroke in Guadeloupe are of type "fast progressor".

We hypothesize that the Afro-Caribbean patients admitted to CHUG for IC would be mostly "fast progressors".

The rate of progression will be determined using brain imaging from the measurement of ischemia volume. This faster progression could be explained by several factors including (1) differences in blood supply between the two populations; (2) environmental and climatic conditions and (3) epigenetic and genetic factors

ELIGIBILITY:
* inclusion criteria:

  * Patients aged 18 and over, admitted for IC due to LVO verified by medical imaging and hospitalized in neurology.
  * Patients residing in Guadeloupe
  * Afro-Caribbean patients: of African ancestry.
  * Emergency inclusion, with exemption from obtaining consent due to the immediate life-threatening emergency situation of the patient (Article L1122-1-3 of the French Public Health Code); as soon as possible, consent to continue will be sought from the patient or, if applicable, from a relative or a trusted person.
  * Patients affiliated to a social security scheme or equivalent
* exclusion criteria:

  * Patients under 18 years old
  * Non-resident patients in Guadeloupe
  * Protected persons (articles L1121-5, L1121-6 and L121-8 of the Public Health Code): pregnant or breastfeeding women, persons deprived of their liberty, under guardianship or curatorship)
  * Withdrawal of consent during the study
  * Patients not affiliated to a social security or equivalent scheme

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with a diagnosis of stroke from LVO identified by medical imaging
Sampling Method: Non-Probability Sample
Enrollment: 135 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2028-01 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
progression of cerebral ischemia of IC in Afro-Caribbean patients admitted to the CHUG with that of patients from Nantes included in the national register ETIS | baseline, day 1,2,3,4 an day 90
  Compare the progression of cerebral ischemia of IC in Afro-Caribbean patients admitted to the CHUG with that of patients from Nantes included in the national register ETIS

SECONDARY OUTCOMES:
Characterizing the profile of Afro-Caribbean patients | baseline
  1. the collateral imaging substitutions in patients of CHUG and CHU de Nantes. The collateral network will be evaluated either by perfusion imaging (Tmax > 6s) or by digitized arterial angiography in a thrombectomy room on the day of stroke according to the ASITN/SIR classification (J0).
Characterizing the profile of Afro-Caribbean patients | baseline
  impact of environmental conditions on ischemia progression rate at Guadeloupe Hospital
Characterizing the profile of Afro-Caribbean | at the end of the suty
  the effect of ischemia-reperfusion induced inflammatory response on ischemia volume

CONTACTS AND LOCATIONS:
Overall Officials: Donald ACCROMBESSI, Doctor, Principal Investigator — CHU de la Guadeloupe; Valérie BASSIEN CASPA, PHD, Study Chair — CHU de la Guadeloupe
Locations (1):
- Centre Hospitalier Universitaire de la Guadeloupe, Pointe-à-Pitre, Guadeloupe, Guadeloupe

IPD SHARING:
Plan to Share IPD: No